CLINICAL TRIAL: NCT03118947
Title: A 52-Week Open-Label Extension Study of Pimavanserin for the Treatment of Agitation and Aggression in Subjects With Alzheimer's Disease
Brief Title: A Study of Pimavanserin for the Treatment of Agitation and Aggression in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-033; 2016-001128-78 (EudraCT Number)
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Agitation and Aggression in Alzheimer's Disease
MeSH Terms: conditions — Psychomotor Agitation | interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pimavanserin 20 mg OR 34 mg per day (Experimental)
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 20 mg, tablet, taken as two 10 mg tablets, once daily by mouth, OR Pimavanserin 34 mg, tablet, taken as two 17 mg tablets, once daily by mouth

SUMMARY:
To evaluate the safety and tolerability of pimavanserin over 52 weeks of treatment in subjects with probable AD who have symptoms of agitation and aggression

ELIGIBILITY:
Inclusion Criteria:

1. Must complete the Week 12 visit in Study ACP-103-032 while continuing to take his/her assigned dose of blinded study drug
2. Can understand the nature of the trial and protocol requirements and provide signed informed consent

   * from patient, if deemed competent to provide consent
   * from an appropriate person (e.g. patient's Legally Authorized Representative (LAR) with the patient's assent) if patient is deemed not competent to provide informed consent.
3. Lives at home or in an assisted living or care facility (but has the capacity to visit the clinic as an outpatient)
4. Has a designated study partner/caregiver who is in contact with the patient at least 3 times a week on 3 separate days
5. Female patients must be of non-childbearing potential or must agree to use an acceptable method of contraception or abstinence, during the study, and 1 month following completion of the study
6. The patient and caregiver are willing and able to participate in all schedule evaluations and complete all required tests

Exclusion Criteria:

1. Patient was significantly non-compliant in Study ACP-103-032
2. The Investigator becomes aware of an impending and unexpected change in the patient's living situation (e.g., change in caregiver, change in facility, moving from home to facility, moving from one family member or caregiver's home to another) that may cause a major disruption in the patient's behavior
3. Patient or study partner/caregiver has a medical condition (e.g., hearing, vision impairments) that would impair the ability to perform the study assessments.
4. Patient is bedridden or has any significant medical condition that is unstable and would place the patient at undue risk from study drug or study procedures
5. Has clinically significant laboratory abnormalities that would jeopardize the safe participation of the patient in the study
6. Has a Global Clinician Assessment of Suicidality (GCAS) score of 3 or 4 based on Investigator's assessment of behavior since the last assessment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (17):
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Neuro-Pain Medical Center, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Pacific Clinical Research Network, San Diego, California
  - Clinical Research Unit, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Quantum Laboratories Inc., Deerfield Beach, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Collier Neurologic Specialists LLC, Naples, Florida
  - Acadia Hospital, Bangor, Maine
  - Alzheimer's Disease Center, Quincy, Massachusetts
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - ANI Neurology, PLLC dba Alzheimer's Memory Center, Charlotte, North Carolina
  - Abington Neurological Associates, Ltd., Willow Grove, Pennsylvania
  - Insite Clinical Research, LLC, DeSoto, Texas
  - Pharmaceutical Research Associates, Inc., Salt Lake City, Utah
- Chile (3):
  - Psicomed Estudios Médicos, Antofagasta
  - Biomedica Research Group, Santiago
  - Especialidades Medicas L y S, Santiago
- CHU de Toulouse - Cite de la sante - Gerontople, Toulouse, Cedex 9, France
- Spain (4):
  - Centro de Atencion Especializada Oroitu, Algorta, Viscaya
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari Mutua de Terrassa, Terrassa
  - Hospital Viamed Montecanal, Zaragoza
- United Kingdom (3):
  - RICE-The Research Institute for the Care of Older People, The RICE Centre, The Royal United Hospital, Bath
  - West London Cognitive Disorders Treatment & Research Unit, Lakeside Mental Health Unit, West Middlesex University Hosp. Site, Isleworth
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label extension study included patients completing double-blind, randomised, placebo-controlled study ACP-103-032 (NCT02992132).
Pre-assignment Details: Patients from parent study ACP-103-032 who were eligible to participate in this study were consented prior to the final procedures performed for study ACP-103-032 at Week 12. The ACP-103-032 Week 12 visit was also considered the baseline visit of study ACP-103-033. The ACP-103-033 result tables are all based on the safety analysis set (n=78).
Groups:
- All Patients: All patients started treatment with pimavanserin 20 mg once daily (QD). At the Week 2 visit, the dose could be increased to 34 mg QD based on the investigator's assessment of clinical response. Subsequently, the dose could be adjusted from 34 mg to 20 mg or from 20 mg to 34 mg at any visit based on clinical response.
Period: Overall Study
Arm/Group | All Patients
Started | 78
Completed | 49
Not Completed | 29
Not completed — Adverse Event | 7
Not completed — Death | 3
Not completed — Lack of Efficacy | 4
Not completed — Non-compliance with study drug | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 3
Not completed — Withdrawal by caregiver | 3
Not completed — Change in patient's living situation | 4
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Treated patients (i.e. patients receiving at least 1 dose of open-label study drug)
Arm/Group | All Patients
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 69
  More than one race | 0
  Unknown or Not Reported | 7
Duration of symptoms of Alzheimer's disease [Mean (Standard Deviation); unit: years] | 6.2 (2.32)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events (TEAEs)
Description: Safety and tolerability of pimavanserin after 52 weeks of treatment in patients with probable Alzheimer's disease who have symptoms of agitation and Aggression, in terms of occurrence of TEAEs
Time Frame: 52 weeks
Population: Treated patients (i.e. patients receiving at least 1 dose of open-label study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 78
Participants | 53

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 3/78
Serious Adverse Events (participants affected / at risk) | 12/78
Other Adverse Events (participants affected / at risk) | 20/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=78)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=78)
Fall (Injury, poisoning and procedural complications) | 7 (7)
Urinary tract infection (Infections and infestations) | 6 (9)
Upper respiratory tract infection (Infections and infestations) | 5 (6)
Agitation (Psychiatric disorders) | 5 (8)
Weight decreased (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03118947/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT03118947/SAP_001.pdf